CLINICAL TRIAL: NCT03661177
Title: Reclaiming Indigenous Food and Health: a Pilot RCT on Health Impacts of Sovereign Nation Diets
Brief Title: Reclaiming Indigenous Food and Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wyoming (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 20180726JK02057
Record Dates: First submitted 2018-09-04; First posted 2018-09-07 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Obesity; Overweight; Diabetes; Hypertension
MeSH Terms: conditions — Obesity; Overweight; Diabetes Mellitus; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diet intervention (Experimental)
  Interventions: Other: Sovereign nation diet
- Control (No Intervention)

INTERVENTIONS:
Other: Sovereign nation diet — We will pilot a RCT with delayed intervention to provisionally assess health impacts of consuming a diet that is 50% indigenous foods for four weeks.
  Other Names: Reclaiming indigenous food and health: a pilot RCT on health impacts of sovereign nation diets
  Arms: Diet intervention

SUMMARY:
The overall purpose of this proposed action-research project is to measure the feasibility of consuming and the impact of indigenous plants and foods on health outcomes among Native American participants.

DETAILED DESCRIPTION:
The overall purpose of this proposed action-research project is to measure the feasibility of consuming and the impact of indigenous plants and foods on health outcomes among Native American participants on the Wind River Indian Reservation (WRIR) in Wyoming.

Participants from the WRIR will be recruited to pilot a randomized control trial (RCT) with a delayed intervention to measure the impacts of consuming a diet that is 50% indigenous foods (based on participant total energy needs and recommended dietary pattern). Specific objectives of the pilot RCT will be to: (1) evaluate the feasibility of access, collection, and consumption of indigenous plants/animals, (2) define precisely what constitutes a "50% indigenous food diet" that will be supplied as the intervention in this trial, (3) quantify the time commitment and logistical challenges to access and collect indigenous foods, (4) evaluate the consumption of indigenous foods on health outcomes including waist circumference, body mass index, blood pressure, blood glucose control, and blood lipid levels, and (5) evaluate the impact of consuming indigenous foods on cultural identity.

The pilot RCT will primarily address objectives 4 and 5. In order to meet these specific objectives, the investigators will pilot a RCT with delayed intervention to provisionally assess health impacts of consuming a diet that is 50% indigenous foods for four weeks. Health outcomes assessed will include biometric measures of waist circumference, body mass index, blood pressure, hemoglobin A1C, total cholesterol with triglycerides; and survey measures of quality of life, cultural identification, and food security.

ELIGIBILITY:
Inclusion Criteria:

* self-identify as living within the boundaries of WRIR (including the city of Riverton)
* self-identify as an enrolled member of the Eastern Shoshone or Shoshone Bannock tribe
* be interested in following a 50% traditional diet for 4 weeks
* 18 years of age or older

Exclusion Criteria:

- Diagnosed with any disorder that causes a compromised immune system (e.g. cancer such as leukemia, HIV/AIDS)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-01-16 (Actual); Primary Completion 2020-03-28 (Actual); Study Completion 2024-06-05 (Actual)

PRIMARY OUTCOMES:
Body mass index | Change in baseline over 5 weeks
  Body mass index (using height and weight) will be measured using a portable stadiometer (to measure height) + Tanita Analyzer (to measure weight). Body mass index parameters for health (i.e. healthy weight is equivalent to a BMI between 18.5-24.9) will be evaluated.
Blood pressure | Change in baseline over 5 weeks
  Both systolic and diastolic pressures will be assessed.
Waist circumference | Change in baseline over 5 weeks
Hemoglobin A1C | Change in baseline over 5 weeks
Lipid panel | Change in baseline over 5 weeks

SECONDARY OUTCOMES:
Mental health change | Change in baseline over 5 weeks
  Measured by 2 statements or questions about general mental health. For each question/statement, participants respond to a 5 point scale (1= none of the time, 5 = all of the time). Statements may be reverse scored for analysis resulting in a higher value indicating a positive change in mental health.
Physical health change | Change in baseline over 5 weeks
  Measured by 12 statements or questions about general health. For each question/statement, participants respond to a 5 point scale (1= none of the time or poor, 5 = all of the time or excellent). A high value on the scale would indicate a positive change in physical health.
Food security change | Change in baseline over 5 weeks
  Measured by 8 statements that people have made about their food situation. For these statements, participants indicate whether the statement was often true, sometimes true, or never true for your household in the last four weeks. Statements will be scored (1=never true, 2 = sometimes true, 3 = often true). Statements may be reverse scored for analysis resulting in a higher value indicating a positive change in food security.
Cultural identity change | Change in baseline over 5 weeks
  Measured by survey questions related to experiences of traditional Native American people. Each item is rated by participants in terms of how much they have participated in each activity (1 = not at all, 7 = a great deal). A high value on the scale would indicate a positive change in cultural identity.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Wyoming, Laramie, Wyoming, United States

IPD SHARING:
Plan to Share IPD: No
PD will be made available to each individual participant, but otherwise only the data summaries will be made available to non-partner parties unless individually arranged and approved by the IRB and project Advisory Board (Restoring Shoshone Ancestral Food Gathering group). The Eastern Shoshone tribe co-owns the data with the research team.